CLINICAL TRIAL: NCT04455542
Title: To Evaluate the Correlation Between Peripheral Neurofilament Levels and Clinical Subtypes of Amyotrophic Lateral Sclerosis and the Severity of Peripheral Motor Axonal Involvement.
Brief Title: Peripheral Neurofilament Levels and Amyotrophic Lateral Sclerosis
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUTH2017198
Record Dates: First submitted 2020-06-28; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Neurofilament levels
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- LMND-ALS: The main clinical manifestations were muscle weakness with atrophy and bundle fibrillation, the pyramidal tract sign was relatively mild, and extensive neurogenic damage with CMAP amplitude decreased could be seen in patients with electromyography.
  Interventions: Other: LMND-ALS
- UMND-ALS: The main clinical manifestations were limb stiffness and spasm, obvious pyramidal tract signs, relatively mild muscle atrophy and fasciculation, and no significant decrease in amplitude of electromyography CMAP.
  Interventions: Other: UMND-ALS
- FAS and FLS: The clinical symptoms were confined to upper limbs (FAS) or lower limbs (FLS) for more than 12 months, and the main manifestations were lower motor neuron involvement signs such as muscle weakness and atrophy
  Interventions: Other: FAS and FLS

INTERVENTIONS:
Other: LMND-ALS — in line with LMND -ALS inclusion criteria, and CMAP amplitude of peripheral motor nerves (CMAP amplitude of the 10 peripheral motor nerves with the most obvious CMAP amplitude decline was selected as the CMAP amplitude for grouping of the patients) was less than the median of CMAP amplitude of LMND -ALS group.
  Groups: LMND-ALS
Other: UMND-ALS — The main clinical manifestations were limb stiffness and spasm, obvious pyramidal tract signs, relatively mild muscle atrophy and fasciculation, and no significant decrease in amplitude of electromyography CMAP.
  Groups: UMND-ALS
Other: FAS and FLS — The clinical symptoms were confined to upper limbs (FAS) or lower limbs (FLS) for more than 12 months, and the main manifestations were lower motor neuron involvement signs such as muscle weakness and atrophy.
  Groups: FAS and FLS

SUMMARY:
To evaluate the correlation between peripheral neurofilament levels and clinical subtypes of amyotrophic lateral sclerosis and the severity of peripheral motor axonal involvement.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a kind of neurodegenerative disease that affects upper and lower motor neurons. In animal model studies have shown that peripheral nerve degeneration in ALS motor function decline, tip peripheral nerve degeneration is of great significance for early progress of ALS may be, at the same time analysis showed that the motor neuron involvement severity and the prognosis of patients with ALS show obvious negative correlation, so finding biomarkers can reflect the motor neuron axonal degeneration is of great significance. Neurofilaments is an intermediate fiber specifically expressed in central and peripheral neurons and can serve as a biomarker for axonal injury, but there is no evidence now that peripheral neurofilament levels have been associated with severity of motor axonal involvement in ALS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lower motor neuron involvement (LMND-ALS), who have visited the Department of Neurology of the Third Hospital of Beijing Medical University since August 2017, meet the diagnostic criteria for ALS in 1998. The main clinical manifestations were muscle weakness with atrophy and bundle fibrillation, the pyramidal tract sign was relatively mild, and extensive neurogenic damage with CMAP amplitude decreased could be seen in patients with electromyography.

  * LMND-ALS CMAP amplitude < median array: in line with LMND -ALS inclusion criteria, and CMAP amplitude of peripheral motor nerves (CMAP amplitude of the 10 peripheral motor nerves with the most obvious CMAP amplitude decline was selected as the CMAP amplitude for grouping of the patients) was less than the median of CMAP amplitude of LMND -ALS group.
  * LMND -ALS CMAP amplitude ≥ median array: meeting LMND -ALS inclusion criteria, and CMAP amplitude of peripheral motor nerves (CMAP amplitude of 10 peripheral motor nerves with the most obvious CMAP amplitude decline was selected as the CMAP amplitude for grouping of the patients) was greater than or equal to the median of CMAP amplitude of LMND -ALS group.
* Patients with upper motor neuron involvement (UMND-ALS): patients with ALS who visited the Department of Neurology of the Third Hospital of Beijing Medical University since August 2017 and met the diagnostic criteria for ALS in 1998. The main clinical manifestations were limb stiffness and spasm, obvious pyramidal tract signs, relatively mild muscle atrophy and fasciculation, and no significant decrease in amplitude of electromyography CMAP.
* Patients with ALS with flail arm syndrome (FAS) and flail leg syndrome (FLS): patients with ALS who met the diagnostic criteria for ALS in 1998 and visited the Department of Neurology of the Third Hospital of Beijing Medical University since August 2017. The clinical symptoms were confined to upper limbs (FAS) or lower limbs (FLS) for more than 12 months, and the main manifestations were lower motor neuron involvement signs such as muscle weakness and atrophy.

Exclusion Criteria:

* Merging other nervous system degenerative diseases (Alzheimer's disease, Parkinson's disease, multiple system atrophy, etc.) to take off the sheath, central nervous system disease, multiple sclerosis, optic myelitis spectrum disorders), peripheral neuropathy (GBS, chronic inflammatory more nerve root sheath sex mental derangement, hereditary peripheral neuropathy, diabetic peripheral neuropathy, vice tumor peripheral neuropathy, secondary to autoimmune diseases ), into the group within a month before the cerebrovascular disease or cerebral or spinal surgery patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lower motor neuron involvement (LMND-ALS), who have visited the Department of Neurology of the Third Hospital of Beijing Medical University since August 2017, meet the diagnostic criteria for ALS in 1998.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
level of neurofilament | 1 year after recruitment
  Venous blood 4 ml was extracted from the three groups of patients for determination of the level of neurofilament.

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, MD.PHD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No